CLINICAL TRIAL: NCT01997008
Title: Optimizing Resilience and Coping in HIV Via Internet Delivery
Acronym: ORCHID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCSF CHR 13-11990
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: HIV Disease; Depression; Affect; Psychological Stress
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Stress, Psychological | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants receive a five week intervention providing the following activities:
  EMA:
  Ecological Momentary Assessment (EMA) of Emotion throughout the day.
  Intervention:
  Positive Events: Participants identify a positive event and then describe how they capitalized on this event.
  Gratitude: Participants identify one more more things that make them feel grateful.
  Mindfulness: Participants participate in a 30 minute guided mindfulness/meditation practice.
  Positive Reappraisal: Participants identify how they reappraised a negative event making it into a positive event.
  Personal Strengths: Participants identify one more more personal strengths. Attainable goals: Participants identify a short-term attainable goal. Participants will outline what they did that day to work toward attaining their week's goal.
  Acts of Kindness: Participants will identify one more more acts of kindness that they engaged in and how it made them feel.
  Interventions: Behavioral: Intervention
- Emotion reporting and EMA notification (No Intervention): Participants report emotions and receive EMA (ecological momentary assessment) text messages on the same regular basis as intervention participants, but receive no interventions.
  EMA detail:
  Ecological Momentary Assessment (EMA) of Emotion throughout the day. We will assess current emotions via email or text message 4 times per day, 2 days per week (one randomly selected week/work day and one randomly selected weekend/non-work day) during the 8 week study period, for a total of 16 days of EMA reporting. Participants will be asked to rate how much they are currently feeling several positive and negative emotions that have been associated with mortality and health: happy, excited, content, appreciative, sad, worried, and fearful.

INTERVENTIONS:
Behavioral: Intervention — Positive Affect Skills Training
  Arms: Intervention

SUMMARY:
This is a feasibility/pilot test of a set of positive affect skills provided online to HIV positive people with elevated depressive symptoms - a Center for Epidemiological Studies Depression Scale D (CES-D) score > 10. The investigators will test the feasibility of recruitment, retention and acceptability of these skills in an online delivery format, determine feasibility and acceptability of daily emotion assessments via text messaging and assess efficacy of these skills for improving psychological well-being this population.

ELIGIBILITY:
Inclusion Criteria:

* HIV +
* 18 or older
* Score of CES-D depression scale >10
* Daily internet access
* Smart phone ownership

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Acceptability of ORCHID content | 5 weeks post enrollment. May be slightly more or less for intervention participants depending on time taken to complete online content.
  We will track participation in both the self-report questionnaires as well as the intervention sessions (e.g., number of ORCHID sessions completed, amount of home practice completed). We will carefully track usage - noting when participants who leave the study drop out to determine if there are particular sessions that are less acceptable than others.
Retention of participants in online delivery format. | 5 weeks post enrollment. May be slightly more or less for intervention participants depending on time taken to complete online content.
  We will track, for each participant who completes a screening questionnaire, where they heard about the study and the proportion who go on to enroll. We will track retention - noting when participants drop out to determine if particular sessions or activities result in less retention than other areas.
Feasibility of an online delivery format. | 5 weeks post enrollment. May be slightly more or less for intervention participants depending on time taken to complete online content.
  We will follow up with participants who have significant missing data to determine areas in which the protocol is feasible and to highlight areas for improvements. We will summarize participant feedback regarding the protocol and will use this feedback to inform the subsequent proposals.

SECONDARY OUTCOMES:
Determine acceptability of multiple daily emotion assessments using text messaging. | 5 weeks post enrollment. May be slightly more or less for intervention participants depending on time taken to complete online content.
  To measure this outcome, we will first document if anyone declines participation due to the perceived burden of the Ecological Momentary Assessment (EMA) protocol. We will carefully document adherence to the protocol and the proportion of assessments that participants complete. In the follow-up interviews, we will have questions specific to the EMA protocol to elicit feedback and suggestions for improvement

OTHER OUTCOMES:
Assess preliminary efficacy of the ORCHID intervention for improving psychological well-being in people living with HIV who have elevated depressive symptoms. | 5 weeks post enrollment. May be slightly more or less for intervention participants depending on time taken to complete online content.
  To address Aim 3 (assess preliminary efficacy of ORCHID on psychological well-being), we will examine means on depression, positive and negative emotion, and perceived stress at each of the assessment points and compare the intervention and emotion reporting only control conditions. Given the small sample size, our analyses will be descriptive and exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Moskowitz, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Moskowitz JT, Hult JR, Duncan LG, Cohn MA, Maurer S, Bussolari C, Acree M. A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test. J Health Psychol. 2012 Jul;17(5):676-92. doi: 10.1177/1359105311425275. Epub 2011 Oct 21. PMID 22021272